CLINICAL TRIAL: NCT06402448
Title: Prevalence of Muscle, Joint and Nerve Pain in Spinal Disorders.
Brief Title: Prevalence of Muscle and Nerve and Joint Pain
Status: Recruiting | Type: Observational
Sponsor: Hadeer Gomaa Ebraheem Aly (Other)
Responsible Party: Sponsor-Investigator, Hadeer Gomaa Ebraheem Aly, physiotherapist, Cairo University
Organization: Cairo University (Other)
Other Study IDs: P.T.REC/012/005032
Record Dates: First submitted 2024-04-19; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Muscle Pain; Joint Pain; Nerve Pain
MeSH Terms: conditions — Myalgia; Arthralgia; Neuralgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: one group containing 300 patients of muscle , joint and nerve pain.
  Interventions: Diagnostic Test: muscle pain , joint pain and nerve pain.

INTERVENTIONS:
Diagnostic Test: muscle pain , joint pain and nerve pain. — to discover the percentage of each tissue that causing pain even it is muscle, joint or nerve in patients with spinal disorders.

SUMMARY:
The purpose of the study is to provide adequate information about the percentage of the main tissue that causing pain in most common spinal disorders either it is muscular, nerve or joint in each spinal parts, that will provide the physical therapist with large data that can be helpful in differential diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. - patients from 18 to 60years
2. - both gender and any condition diagnosed by orthopedic physician with spinal disorders
3. - pre and post operative patient may be included.

Exclusion Criteria:

1. viscerogenic pain
2. cancer
3. psychogenic pain or psychogenic disorder
4. rheumatoid arthritis
5. fibromyalgia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients from 18 to 6o years , both gender and any condition diagnosed by orthopedic physician with spinal disorders and pre and post operative patient may be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
muscle pain | 5 months
  muscle pain with pressure algometer ,stretch and resisted range of motion .
joint pain | 5 months
  joint pain with joint play and physiological range of motion .
nerve pain | 5 months
  nerve pain with tinel sign and neural tension test .

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Egypt